CLINICAL TRIAL: NCT06691347
Title: Towards Evidence-based PTSD Care in Norwegian Specialist Health Services - A Randomized Controlled Trial
Brief Title: Effectiveness of Trauma Treatment in the Specialist Health Care Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 716204
Record Dates: First submitted 2024-09-26; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Post Traumatic Stress Disorder PTSD; Quality of Life; Functional Outcome; Complex Post-Traumatic Stress Disorder; Eye Movement Desensitization and Reprocessing; Cognitive Therapy
MeSH Terms: conditions — Combat Disorders | interventions — Eye Movement Desensitization Reprocessing; Cognitive Behavioral Therapy

STUDY DESIGN:
Masking Description: The Investigator will be blinded to the random allocation of patients, but will have knowledge of the interventions when treatment begins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Movement Desensitization and Reprocessing (Experimental): Patients will receive EMDR as their main treatment method of PTSD. EMDR processes trauma memories while engaging in bilateral stimulation to help rewire the brain's response to trauma and decrease emotional distress.
  Interventions: Behavioral: Eye movement desensitization and reprocessing
- Cognitive Therapy for PTSD (Experimental): Patients will receive CT-PTSD as their main treatment method of PTSD. CT-PTSD focuses on techniques such as cognitive restructuring and exposure therapy to help individuals reframe trauma and reduce intrusive memories and emotional distress.
  Interventions: Behavioral: Cognitive therapy for PTSD

INTERVENTIONS:
Behavioral: Eye movement desensitization and reprocessing — Psychotherapy with EMDR. A therapist guides the client in recalling distressing events while simultaneously following a stimulus, like a moving light or tapping. The idea is that this bilateral stimulation helps reduce the intensity of the traumatic memory, allowing clients to gain perspective and lessen emotional distress associated with it. The standard treatment protocol includes up to 24 weekly sessions.
  Other Names: EMDR
  Arms: Eye Movement Desensitization and Reprocessing
Behavioral: Cognitive therapy for PTSD — Psychotherapy with CT-PTSD. A therapist works with the client to understand how they interpret their trauma and identify distorted thinking patterns that fuel their PTSD symptoms. Through guided discussions, written exercises, and sometimes "re-living" the trauma in a controlled way, clients learn to reshape these beliefs, gain a more balanced perspective, and reduce symptoms like hypervigilance, flashbacks, and avoidance behaviors. The standard treatment protocol includes up to 24 weekly sessions.
  Other Names: CT-PTSD
  Arms: Cognitive Therapy for PTSD

SUMMARY:
Post-traumatic stress disorder (PTSD) is a common mental illness. Treatments for PTSD are regarded as highly effective, but a large-scale, prospective, longitudinal randomized controlled trial comparing the effectiveness of these treatments has been requested by the research community. This study aims to conduct a comprehensive investigation into the effectiveness of two prominent PTSD therapies, eye movement desensitization and reprocessing (EMDR) and cognitive therapy for PTSD (CT-PTSD), within the Norwegian specialist health care services. The study aims to compare the therapy effectiveness, including their impact on comorbid disorders, complex PTSD symptoms, and functional outcomes post-treatment. Patients will be randomly assigned to EMDR or CT-PTSD and given manualized therapy aligned with their treatment goals. Each arm aims to recruit 135 patients, resulting in a total sample size of 270 patients.

The main objective of this study is to examine the growth curves of the two methods and how patient characteristics affect their developments. Secondary short-term aims include (1) investigating the impact of EMDR and CT-PTSD on complex PTSD symptoms, (2) assessing effects on other clinical conditions and functional outcomes, and (3) exploring whether the therapeutic alliance mediates treatment effects. Secondary long-term aims are (1) to assess the long-term effects of EMDR and CT-PTSD on PTSD symptoms and (2) to explore the impact of extended or additional treatments on outcomes.

DETAILED DESCRIPTION:
Participants will be recruited from Asker DPS, Bærum DPS, Drammen DPS, and Ringerike DPS. They were referred to DPS for PTSD treatment, either by general practitioners, other primary health care services in their municipality, or psychiatric hospitals. This study is a longitudinal multi-assessment 2-arm RCT and does not include a treatment as usual group. The standard treatment protocol includes up to 24 weekly sessions. Conversely, if no discernible improvement is seen after 10 sessions, it is recommended to terminate treatment. The clinical assessment consists of self-administered questionnaires collected through CheckWare, which is a digital platform developed for healthcare services. They will be asked to report symptoms of PTSD, depression, anxiety, psychosis, alcohol/drug use, functional outcomes, working alliance. Before treatment starts, patients will complete baseline assessments. Throughout the treatment phase, all patients will be requested to fill out self-administered questionnaires after each session.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* meeting criteria for PTSD based on the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) with a total score ≥23

Exclusion Criteria:

* insufficient mastery of the Norwegian language
* severe intellectual impairment (estimated IQ of 70 or less)
* comorbid psychiatric illnesses in an acute phase where other types of treatment need to be prioritized (e.g. hospitalization)
* history of EMDR or CT-PTSD treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Changes in PTSD-symptoms | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in PTSD checklist for DSM-V (PCL-5) scores. The PCL-5 consists of 20 items on a 5-point Likert scale ranging from 0-4. Total scores range from 0-80, where a higher score signifies a worse outcome.
Changes in PTSD-symptoms | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  The International trauma questionnaire (ITQ) scores. The ITQ consists of 18 items on a 5-point Likert scale ranging from 0-4. Total scores range from 0-72, where a higher score signifies a worse outcome.

SECONDARY OUTCOMES:
Changes in comorbid illnesses | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in symptoms related to depression as measured with The Beck Depression Inventory-II (BDI). The BDI-II consists of 21 items on a 4-point Likert scale ranging from 0-3. Total scores range from 0-63, where a higher score signifies a worse outcome.
Changes in comorbid illnesses | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in symptoms related to anxiety as measured with The Beck Anxiety Inventory (BAI). The BAI consists of 21 items on a 4-point Likert scale ranging from 0-3. Total scores range from 0-63, where a higher score signifies a worse outcome.
Changes in comorbid illnesses | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in symptoms related to psychosis as measured with MULVARP. MULVARP consists of Prodromal Questionnaire (PQ-16). It consists of 16 items on a 4-point Likert scale ranging from 0-3. Total scores range from 0-48, where a higher score signifies a worse outcome.
Changes in comorbid illnesses | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in symptoms related to alcohol use as measured with Alcohol Use Disorders Identification Test (AUDIT). The AUDIT consists of 10 items on a 5-point Likert scale ranging from 0-4, with the exception of questions 9 and 10 which have possible responses of 0, 2 and 4. Total scores range from 0-40, where a higher score signifies a worse outcome.
Changes in comorbid illnesses | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in symptoms related to drug use as measured with Drug Use Disorders Identification Test (DUDIT). The DUDIT consists of 11 items on a 5-point Likert scale ranging from 0-4, with the exception of questions 9 and 10 which have possible responses of 0, 2 and 4. Total scores range from 0-44, where a higher score signifies a worse outcome.
Changes in functional outcomes | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in Quality of Life questionnaire (QoL10) scores. The QoL10 consists of 10 items on a 5-point Likert scale ranging from 1-5. Total scores range from 0-50, where a higher score signifies a worse outcome.
Changes in functional outcomes | From enrollment to the end of treatment at 24 weeks. Follow up at 3, 6 and 12 months
  Changes in Work and Social Functioning (WSAS) scores. The WSAS consists of 5 items on a 9-point Likert scale ranging from 0-8. Total scores range from 0-40, where a higher score signifies a worse outcome.

OTHER OUTCOMES:
The impact of therapeutic alliance on treatment effectiveness | From enrollment to the end of treatment at 24 weeks
  Changes in Working Alliance Inventory scores will be used to evaluate the interventions. The WAI consists of 16 items on a 5-point Likert scale ranging from 1-5. Total scores range from 16-80, where a higher score signifies a better alliance.
In case of re-referral: number of days until re-referral | From end of treatment to 12 months afterwards
  Total number of days from the end of treatment until patients are re-referred to the clinics within the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Susie Fu, Ph.D, Cand. Psychol., Principal Investigator — Vestre Viken Health trust
Locations (1):
- Vestre Viken Health Trust, Drammen, Akershus, Norway

IPD SHARING:
Plan to Share IPD: No